CLINICAL TRIAL: NCT06223659
Title: Investigating the Use of EMLA Topical Cream for Patients Receiving Intra-Dermal Technetium 99 Injections for Lymphoscintigraphy for Cutaneous Cancers
Brief Title: EMLA Topical Cream for Treatment of Pain in Patients Receiving Intra-Dermal Technetium 99 Injections for Lymphoscintigraphy for Skin Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Carlo Contreras, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OSU-23046; NCI-2023-10465 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-01-02; First posted 2024-01-25 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-01

CONDITIONS: Cutaneous Melanoma; Merkel Cell Carcinoma; Skin Squamous Cell Carcinoma
MeSH Terms: conditions — Melanoma; Carcinoma, Merkel Cell | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 2 (placebo cream) (Placebo Comparator): Patients apply placebo cream topically to skin 30 minutes prior to Tc99 lymphoscintigraphy procedure.
  Interventions: Drug: Placebo Administration; Other: Questionnaire Administration
- Cohort 1 (EMLA cream) (Experimental): Patients apply EMLA cream topically to skin 30 minutes prior to Tc99 lymphoscintigraphy procedure.
  Interventions: Drug: Eutectic Mixture of Local Anesthetics; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Eutectic Mixture of Local Anesthetics — Apply topically to skin
  Other Names: EMLA; Lidocaine-Prilocaine Eutectic Mixture; Lidocaine/Prilocaine; Oraqix
  Arms: Cohort 1 (EMLA cream)
Drug: Placebo Administration — Apply topically to skin
  Arms: Cohort 2 (placebo cream)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests how well EMLA topical cream works in treating pain in patients with skin cancers receiving Technetium 99 injections for a lymphoscintigraphy mapping procedure. A lymphoscintigraphy mapping procedure is used to find the main or lead lymph node (tissue that fight infection) so it can be removed and checked for tumor cells. Using lymphoscintigraphy to highlight and then surgically remove lymph nodes is standard way to treat skin cancer for many patients. The Technetium 99 injections used for lymphoscintigraphy can be briefly painful due to the sensitivity of the nerve endings in the skin. The EMLA topical cream, which contains a numbing medicine to block pain from nerve endings, has been studied in breast cancer patients with a difference in pain reported, but this is the first time it has been studied in patients undergoing lymphoscintigraphy for skin cancer. This study may help researchers learn whether the use of EMLA cream may improve the associated pain at the time of the lymphoscintigraphy procedure.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate if the application of eutectic mixture of local anesthetics (EMLA) topical cream (2.5% lidocaine mixed with 2.5% prilocaine) prior to intra-dermal Technetium 99 sulfur colloid (Tc99 injection) for lymphoscintigraphy can improve associated pain.

OUTLINE: Patients are randomized to 1 of 2 cohorts.

COHORT 1: Patients apply EMLA cream topically to skin 30 minutes prior to Tc99 lymphoscintigraphy procedure.

COHORT 2: Patients apply placebo cream topically to skin 30 minutes prior to Tc99 lymphoscintigraphy procedure.

ELIGIBILITY:
Inclusion Criteria:

* Biologic males or females
* 18 - 99 years of age
* Histologically confirmed cutaneous melanoma, Merkel cell carcinoma, squamous cell carcinoma, or other cutaneous malignancy for which lymphoscintigraphy and sentinel lymph node biopsy has been recommended.

Exclusion Criteria:

* Known allergy or intolerance to EMLA cream, lidocaine, prilocaine, or any other local anesthetic
* History of adhesive allergy
* Contraindication to Tc99 injection for sentinel lymph node mapping
* Incarcerated patients
* Patients incapable of independently providing consent
* Mucosal or genital lymphoscintigraphy site
* Pregnancy
* Participant self-declared or Ohio State University (OSU) medical chart listing chronic pain as a pre-existing diagnosis
* Participants with chronic pain as defined by the Centers for Disease Control and Prevention (CDC):"pain lasting 3 months or more that can be caused by a disease or condition, injury, medical treatment, or unknown reason" excluding those with stable co-morbid conditions such as peripheral neuropathy, fibromyalgia, arthritis, and cancer-related pain who do not require narcotics. Patients who require narcotics at any time within the 7-day period leading up to the procedure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score | Up to 1 year
  Pain will be measured on a Defense and Veterans Pain Rating 10-point scale where 1 is the lowest measure of pain, and 10 is the highest pain. Will be analyzed using an independent samples t-test to compare the mean pain score of the two cohorts. Descriptive statistics of patient demographics and adverse events will also be reported.

SECONDARY OUTCOMES:
Incidence of adverse events | 30 minutes after lymphoscintigraphy injection
  Reported side effects will be recorded and compared between the two groups using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo M Contreras, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu